CLINICAL TRIAL: NCT04266665
Title: Effect of Dexmedetomidine on Brain Homeostasis and Neurocognitive Outcome of Patients Undergoing Brain Tumor Exclusion
Brief Title: Effect of Dexmedetomidine on Brain Homeostasis and Neurocognitive Outcome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Georgia Tsaousi (Other)
Responsible Party: Sponsor-Investigator, Georgia Tsaousi, Assistant Professor, Aristotle University Of Thessaloniki
Organization: Aristotle University Of Thessaloniki (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DexProB
Record Dates: First submitted 2020-02-02; First posted 2020-02-12 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Brain Tumor; Metabolic Disturbance; Inflammatory Response; Oxygen Deficiency
Keywords: dexmedetomidine; brain oxygenation; biomarkers; neuroinflammation; brain metabolism; neurocognitive outcome
MeSH Terms: conditions — Brain Neoplasms; Hypoxia; Neuroinflammatory Diseases | interventions — Dexmedetomidine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Active Comparator): Dexmedetomidine 2 μg/ml will be given as bolus 1mg/kg for 10 minutes with a maintenance dose of 0.8μg/kg/h until surgery completion
  Interventions: Drug: Dexmedetomidine
- Normal saline (Placebo Comparator): Normal saline (NaCl 0.9%) administration will start 10 minutes after anesthesia induction and maintained throughout the surgical procedure.
  Interventions: Other: Normal saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine 2 μg/ml will be given as bolus 1mg/kg for 10 minutes with a maintenance dose of 0.8μg/kg/h until surgery completion
  Other Names: Dexdor
  Arms: Dexmedetomidine
Other: Normal saline — Equivalent doses for a solution containing 2mcg/ml of the tested drug calculating for a bolus 1mg/kg for 10 minutes with a maintenance dose of 0.8μg/kg/h until surgery completion
  Other Names: NaCl 0.9%
  Arms: Normal saline

SUMMARY:
Brain tumor surgery is commonly associated with different degrees of preoperative intracranial hypertension and surrounding tumor edema, elicited by tumor underlying pathophysiology. During craniotomy for brain tumor resection maintenance of hemodynamic stability and intracranial homoeostasis is of paramount importance. Disordered hemodynamics or adverse stress may activate the immune inflammation or neuroendocrine responses and lead to a surge of inflammatory mediators and stress hormones, which are implicated in secondary brain insults.

Adverse physiological responses caused by intraoperative disordered hemodynamics or surgery-related damage, may lead to some secondary brain injury (such as cerebral edema or cerebral hemorrhage), aggravating damage to brain tissue and affecting the recovery from anesthesia, cognition and prognosis in patients.

Prevention of secondary brain injury is a key-endpoint to improve clinical outcomes in glioma patients undergoing craniotomy.

Alpha2-adrenoceptor agonists have been widely used for sedation, analgesia and anti-sympathetic actions for many years, but the definite evidence of their potential use as neuroprotectants has so far been confined to animal studies, yet the findings are inconsistent.

Dexmedetomidine (DEX) has been demonstrated to be a new type a2 adrenergic receptor (a2-AR) agonist, which can selectively bind with the a1 and a2 adrenergic receptor, and playing a dual role by restraining the activity of sympathetic nervous and stimulating the vagus nerve. Dexmedetomidine (DEX) also plays an important role in in inhibiting inflammatory and neuroendocrine responses. Animal experiments showed that the right must have a dexmedetomidine neuro-protective effect. However, the brain-protective effect of dexmedetomidine in anesthesia of craniotomy resection of glioma has not been reported.

Thus, the aim of this study was to explore the effect of dexmedetomidine on perioperative brain protection, as well as cerebral oxygenation and metabolic status aiming to provide a basis for clinical rational drug use in patients undergoing craniotomy resection of glioma.

DETAILED DESCRIPTION:
Each participant will receive standard monitoring (ECG, SpO2, SBP, BIS, urine output, temperature). More detailed hemodynamic monitoring will be obtained by Edwards Lifesciences ClearSight system (CO, CI, SV, SVI, SVV, SVR, SVRI).

TCI Propofol and Remifentanil will be the agents of choice for induction and maintenance in anesthesia and cisatracurium will be used for neuromuscular blockade for intubation.

Protective mechanical ventilation will be chosen (7ml/kg IBW) with a respiratory rate to obtain a PaCO2 of 35-40 mmHg. PEEP will be changed for the best PaO2/FiO2 ratio and FiO2 of choice will be 0.5.

The radial artery catheterization will be applied for direct blood pressure measurement and arterial blood gas sampling (pH, PaO2, PaCO2, HCO3, BE, osmolality, lactic acid, Hb, glucose, Na and K will be measured).

The jugular bulb ipsilateral to the craniotomy site will be catheterized for receiving blood samples for blood gas analysis. The following oxygenation and metabolic parameters / derivates will be measured or calculated: SjvO2, pH, PjvO2, PjvCO2, HCO3, BE, Osmolality, Lactic acid jv, Hb, Glucose, Na, K, AjvDO2, AjvCO2, O2ERbr, eRQbr, AjvDL, and LOI.

Dexmedetomidine or normal saline (placebo) administration will start 10 minutes after anesthesia induction and maintained throughout the surgical procedure.

Phases

* T0: 5 minutes before administration of either DEX or placebo
* T15: 10 minutes after administration of either DEX or placebo
* T30: 30 minutes after administration of either DEX or placebo
* T60: 60 minutes after administration of either DEX or placebo
* T120: 120 minutes after administration of either DEX or placebo
* T240: 240 minutes after administration of either DEX or placebo
* End of surgical procedure Blood samples for measuring S-100b, NSE, cortisol, TNF-a and IL-6 will be obtained at phases T0, end of surgery and 24 hours after administration of either DEX or placebo.

Neurocognitive testing will be performed before surgery, 1 week and 1 month later using Karnofsky Performance Status (KFS), Mini Mental State Exam (MMSE), Μontreal Cognitive Assessment (MoCA) and Addenbrooke's Cognitive Exam (ACE III).

Intraoperative consumption of propofol and remifentanil will also be recorded

ELIGIBILITY:
Inclusion Criteria:

* ASA-PS 1-3 (American Society of Anesthesiologists Physical Status classification)
* Scheduled for elective or semi-elective craniotomy for brain tumor resection
* Signed informed consent

Exclusion Criteria:

* History of craniotomy at the same site
* Morbid obesity
* Delirious person before surgery
* Preoperative heart rate (HR) <45 beats/min or second or third degree AV block
* Treatment with a-methyldopa, clonidine or other a2-adrenergic agonist
* Pregnancy
* Liver or renal failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2020-03-12 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Changes in S-100b protein | End of surgical procedure and 24 hours postoperatively
  Alterations in S-100b (μg/L) after intravenous infusion of equivalent doses of dexmedetomidine or placebo (normal saline)
Changes in NSE | End of surgical procedure and 24 hours postoperatively
  Alterations in NSE (ng/ml) after intravenous infusion of equivalent doses of dexmedetomidine or placebo (normal saline)

SECONDARY OUTCOMES:
Changes in serum cortisol | End of surgical procedure and 24 hours postoperatively
  Alterations in serum cortisol (μg/dl) levels after intravenous infusion of equivalent doses of dexmedetomidine or placebo (normal saline)
Changes in serum TNF-a | End of surgical procedure and 24 hours postoperatively
  Alterations in serum TNF-a (pg/ml) levels after intravenous infusion of equivalent doses of dexmedetomidine or placebo (normal saline)
Changes in serum IL-6 | End of surgical procedure and 24 hours postoperatively
  Alterations in serum IL-6 (pg/ml) levels after intravenous infusion of equivalent doses of dexmedetomidine or placebo (normal saline)
Changes in Mini-Mental State Exam (MMSE) | 1 week and 1 month after the end of surgical procedure
  Alterations in Mini-Mental State Exam (MMSE) after intravenous infusion of equivalent doses of dexmedetomidine or placebo (normal saline)
Changes in Μontreal Cognitive Assessment (MoCA) | 1 week and 1 month after the end of surgical procedure
  Alterations in Μontreal Cognitive Assessment (MoCA) after intravenous infusion of equivalent doses of dexmedetomidine or placebo (normal saline)
Changes in Addenbrooke's Cognitive Exam (ACE III) | 1 week and 1 month after the end of surgical procedure
  Alterations in Addenbrooke's Cognitive Exam (ACE III) after intravenous infusion of equivalent doses of dexmedetomidine or placebo (normal saline)

OTHER OUTCOMES:
Changes in jugular venous oxygen saturation | 10, 30, 60, 120, 240 minutes after commencing the infusion of the tested agent and end of surgical procedure
  Alterations in jugular venous oxygen saturation (%), after intravenous infusion of equivalent doses of dexmedetomidine or placebo (normal saline)
Changes in arterio-jugular oxygen difference (AjvDO2) | 10, 30, 60, 120, 240 minutes after commencing the infusion of the tested agent and end of surgical procedure
  Alterations in arterio-jugular oxygen difference (AjvDO2 [ml/dl]), after intravenous infusion of equivalent doses of dexmedetomidine or placebo (normal saline)
Changes in arterio-jugular carbon dioxide difference (AjvCO2) | 10, 30, 60, 120, 240 minutes after commencing the infusion of the tested agent and end of surgical procedure
  Alterations in arterio-jugular carbon dioxide difference (AjvCO2 [mmHg]), after intravenous infusion of equivalent doses of dexmedetomidine or placebo (normal saline)
Changes in brain oxygen extraction ratio (O2Erbr) | 10, 30, 60, 120, 240 minutes after commencing the infusion of the tested agent and end of surgical procedure
  Alterations in brain oxygen extraction ratio (O2Erbr [%]), after intravenous infusion of equivalent doses of dexmedetomidine or placebo (normal saline)

CONTACTS AND LOCATIONS:
Overall Officials: Georgia Tsaousi, Professor, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No